CLINICAL TRIAL: NCT05013814
Title: Comparison of the Tactile Functions and the Effects of Possible Tactile Deficit on Motor Function in Unilateral Cerebral Palsy and the Typically Developed Children
Brief Title: The Effect of Tactile Deficit on Motor Function in Unilateral Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.312
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy; Rehabilitation; Tactile Perception
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with unilateral cerebral palsy
  Interventions: Diagnostic Test: Semmes-Weinstein monofilament test; Diagnostic Test: Box and Block Test; Diagnostic Test: 9-Hole Peg Test; Diagnostic Test: Duruöz Hand Index (DHI); Diagnostic Test: Jamar hand dynamometer; Diagnostic Test: Hydraulic pinch gauge
- Typically developed children
  Interventions: Diagnostic Test: Semmes-Weinstein monofilament test; Diagnostic Test: Box and Block Test; Diagnostic Test: 9-Hole Peg Test; Diagnostic Test: Duruöz Hand Index (DHI); Diagnostic Test: Jamar hand dynamometer; Diagnostic Test: Hydraulic pinch gauge

INTERVENTIONS:
Diagnostic Test: Semmes-Weinstein monofilament test — Tactile function was evaluated mainly as tactile registration by using 20-item Semmes-Weinstein monofilament (SWM) kit. The monofilament was applied three times with a pseudorandom order to distal pad of the thumb, index, 4th and 5th digits (C6, C7 and C8 dermatomes). The lowest value of monofilament was recorded which the child was able to correctly identify at least one touch out of three
Diagnostic Test: Box and Block Test — Box and Block Test (BBT) was used for dexterity assessment. The BBT measures unilateral gross manual dexterity. The child was asked to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size within 60 seconds
Diagnostic Test: 9-Hole Peg Test — 9-Hole Peg Test (9-HPT) is used to measure finger dexterity. Firstly, the child takes the pegs from a container, one by one, and place them in the holes on the board; then participant removes the pegs from the holes and replaces them back into the container. The total time taken to complete the test is recorded in seconds.
Diagnostic Test: Duruöz Hand Index (DHI) — Duruöz Hand Index (DHI) is an 18-item self-report questionnaire regarding ability to carry out manual tasks. Individual items are scored on a 6-point Likert scale where 0=without difficulty and 5=impossible. The total score ranges from 0-90 with higher scores indicating poorer hand function.
Diagnostic Test: Jamar hand dynamometer — Hand grip strength was measured by using Jamar hydraulic hand dynamometer. Measurement was done with the participant in sitting position and the elbow at 90 degrees of flexion. The force has most commonly been measured in kilograms according to the amount of static force that the hand can squeeze around the dynamometer.
Diagnostic Test: Hydraulic pinch gauge — Hydraulic pinch gauge is used for evaluation of finger grip strength. The evaluation method was the same as Jamar hand dynamometer.

SUMMARY:
Cerebral palsy(CP) is the most common cause of disability in childhood. The motor spectrum of disorders is characterized by abnormal muscle tone, posture, and movement. The motor disorders of CP are often accompanied by disturbances of sensation, perception, cognition and behavior. Besides classical appearance of symptomatology, tactile impairment takes an important place to be evaluated. Assessment of the integrity of tactile function composes of two main steps: tactile registration and tactile perception. Our main goal is the define the effect of tactile impairment on hand motor function with the usage of identical assessment tools in patients with unilateral cerebral palsy (UCP) and typically developed children (TDC).

ELIGIBILITY:
Inclusion Criteria:

* Ages between 5-15 years
* Being evaluated as Class I-II-III in Gross Motor Function Classification System
* Being evaluated as Class I-II-III in Manual Ability Classification System

Exclusion Criteria:

* Inability to understand and/or follow test instructions due to intellectual or behavioral difficulties
* History of upper extremity botulinum toxin type A injection in the last three months,
* Previous upper extremity orthopedic surgery
* History of major trauma, and visual impairment

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of 2 groups. In the group of typically developed children, there are healthy children who do not have a disease that will affect normal development. The other group includes children diagnosed with unilateral cerebral palsy.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with tactile dysfunction in both groups | 1 day (Single time point)
  Comparison of the number of patients with tactile dysfunction according to the Semmes-Weinstein monofilament test scores.
Mean score of gross manual dexterity assessment test in all participants | 1 day (Single time point)
  Mean score of Box-Block Test was used to compare gross manual dexterity assessment in both groups
Mean score of hand grip strength test in all participants | 1 day (Single time point)
  Mean score of Jamar dynamometer measures was used to compare hand grip strength in both groups
Mean score of hand function test in all participants | 1 day (Single time point)
  Mean score of Duruöz Hand Index was used to compare hand function in both groups
Mean score of finger dexterity assessment test in all participants | 1 day (Single time point)
  Mean score of 9-Hole Peg Test was used to compare finger dexterity assessment in both groups
Mean score of finger grip strength test in all participants | 1 day (Single time point)
  Mean score of pinch gauge measures was used to compare finger grip strength in both groups

SECONDARY OUTCOMES:
Mean score of gross manual dexterity assessment test according to the tactile function | 1 day (Single time point)
  Tactile function was determined by the Semmes-Weinstein monofilament score. The Box-Block Test scores were compared between those with normal and impaired tactile function in the unilateral cerebral palsy group.
Mean score of hand grip strength test according to the tactile function | 1 day (Single time point)
  Tactile function was determined by the Semmes-Weinstein monofilament score. The Jamar dynamometer scores were compared between those with normal and impaired tactile function in the unilateral cerebral palsy group.
Mean score of finger grip strength test according to the tactile function | 1 day (Single time point)
  Tactile function was determined by the Semmes-Weinstein monofilament score. The pinch gauge scores were compared between those with normal and impaired tactile function in the unilateral cerebral palsy group.
Mean score of hand function test according to the tactile function | 1 day (Single time point)
  Tactile function was determined by the Semmes-Weinstein monofilament score. The Duruöz Hand Index scores were compared between those with normal and impaired tactile function in the unilateral cerebral palsy group.
Mean score of finger dexterity assessment test according to the tactile function | 1 day (Single time point)
  Tactile function was determined by the Semmes-Weinstein monofilament score. The 9-Hole Peg Test scores were compared between those with normal and impaired tactile function in the unilateral cerebral palsy group.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag-Saygi, MD, Study Director — Marmara University
Locations (1):
- Marmara University Pendik Education and Research Hospital, Istanbul, Turkey (Türkiye)